CLINICAL TRIAL: NCT00856973
Title: A Randomized, Placebo Controlled, Double Blind, Fixed Dose Study of the Efficacy and Safety of Eszopiclone in Children (6 to 11 Years) and Adolescents (12 to 17 Years) With Attention Deficit/Hyperactivity Disorder Associated Insomnia
Brief Title: Safety & Efficacy Study of Study Drug (Eszopiclone) in Children and Adolescents With Attention-deficit/Hyperactivity Disorder - Associated Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-246
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-05

CONDITIONS: Insomnia; Attention Deficit Hyperactivity Disorder
Keywords: Hypnotic; Eszopiclone; Attention Deficit/Hyperactivity Disorder; Insomnia; Children; Adolescent; Polysomnography; Actigraphy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose eszopiclone (Experimental): 1 mg eszopiclone for 6-11 years, 2 mg for 12-17 years
  Interventions: Drug: eszopiclone
- High dose eszopiclone (Experimental): 2 mg eszopiclone for 6-11 years, 3 mg eszopiclone for 12-17 years
  Interventions: Drug: eszopiclone
- Placebo (Placebo Comparator): Placebo 6-17 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eszopiclone — 1 mg eszopiclone for 6-11 years, 2 mg for 12-17 years
  Arms: Low dose eszopiclone
Drug: eszopiclone — 2 mg eszopiclone for 6-11 years, 3 mg eszopiclone for 12-17 years
  Arms: High dose eszopiclone
Drug: Placebo — 1 tablet per day for 12 weeks
  Arms: Placebo

SUMMARY:
A multi center, randomized study to evaluate the efficacy and safety of eszopiclone compared to placebo in children (6-11 years of age, inclusive) and adolescents (12-17 years of age, inclusive) with attention deficit/hyperactivity disorder (ADHD) associated insomnia.

DETAILED DESCRIPTION:
This is a multi center, randomized, double blind, placebo controlled, fixed dose study of eszopiclone in pediatric subjects 6-17 years of age, inclusive, with ADHD associated insomnia. Subjects will be randomized at approximately 1:1:1 to either low dose oral eszopiclone (1 mg for children ages 6-11 years, 2 mg for adolescents ages 12-17 years), high dose oral eszopiclone (2 mg for children ages 6-11 years, 3 mg for adolescents ages 12-17 years) or placebo. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female 6 to 17 years of age, inclusive, at the time of consent.
* Subject must have a diagnosis of ADHD as defined by DSM-IV criteria
* Subject must have documented ADHD associated insomnia, defined as the subject or subject's parent/legal guardian having reported repeated difficulty with sleep initiation (sleep latency >30 minutes) or consolidation, (wake time after sleep onset >45 minutes) despite adequate age appropriate time and opportunity for sleep.
* Subject's Baseline PSG must reveal either >30 minutes latency to persistent sleep (LPS) or >45 minutes wake after sleep onset (WASO).
* Subject or subject's parent/legal guardian should have reported daytime functional impairment as a result of sleep problems.
* Subject or subject's parent/legal guardian should have reported attempted and failed behavioral interventions for sleep problems, including a regular bedtime and rise time
* Subject's sleep disturbance must not be attributable to either the direct physiologic effect of a drug of abuse or misuse of a prescribed medication whether it is being used as intended or in an illicit manner.(Female subjects ≥8 years of age must have a negative serum pregnancy test)
* Subject must be in general good health
* Subject must be able to swallow tablets.
* If subject is currently taking medication for ADHD, they must be on a stable dose and regimen for a minimum of 1 month prior to the time of consent

Exclusion Criteria:

* Subject with weight <10th percentile for age and gender
* Subject has any clinically significant or unstable medical illness/abnormality or chronic disease.
* Subject has a documented history of Bipolar I or II Disorder, major depression, conduct disorder, generalized anxiety disorder or any history of psychosis.
* Subject has periodic limb movement >5 times per hour, as demonstrated on Baseline PSG.
* Subject has sleep disordered breathing, as demonstrated on Baseline PSG.
* Subject has another primary sleep disorder, a secondary sleep disorder, or any other known or suspected medical or psychiatric condition that has affected or may affect sleep
* Subject has a history of circadian rhythm disorder or will travel across ≥3 time zones more than once during the study.
* Subject has organic brain disease, or a history of febrile seizures.
* Subject is, in the opinion of the investigator, at suicidal or homicidal risk.
* Female subject who is pregnant or lactating or planning to become pregnant.
* Subject has taken any psychotropic medication without an appropriate washout period (≥5 half-lives) prior to randomization.
* Subject has a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions.
* Subject has a history of allergic reaction or has a known or suspected sensitivity to racemic zopiclone, eszopiclone, or any substance that is contained in the formulation.
* Subject has a history of alcohol or substance abuse within 3 months of study participation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 486 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (73):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Dothan Behavioral Medicine Clinic, Dothan, Alabama
  - Metropolitan Neuro Behavioral Institute, Chandler, Arizona
  - PsyPharma Clinical Research, Phoenix, Arizona
  - REM Medical Clinical Research, Tucson, Arizona
  - Paul E. Wylie, Little Rock, Arkansas
  - AV Institute, Inc., Carson, California
  - Clinical Innovations, Inc., Costa Mesa, California
  - Avastra Clinical Trials, Fountain Valley, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Pacific Institute for Medical Research Inc, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - North County Clinical Research (NCCR), Oceanside, California
  - Pacific Clinical Research Medical Group, Orange, California
  - SDS Clinical Trials, Orange, California
  - California Clinical Trials Medical Group, Paramount, California
  - Clinical Innovations, Inc., Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Clinical Innovations, Inc., San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Clinical Innovations, Inc., Santa Ana, California
  - Elite Clinical Trials, Wildomar, California
  - Delta Waves, INC, Colorado Springs, Colorado
  - Sarkis Clinical Trials, Gainesville, Florida
  - MD Clinical, Hallandale, Florida
  - Florida Clinical Research Center LLC, Maitland, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - SomnoMedics, LLC, Tampa, Florida
  - Pediatric Epilepsy and Neurology Specialists, Tampa, Florida
  - Neuro Trials Research, Inc., Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Mountain West Clinical Trials, Eagle, Idaho
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - AMR Baber Research Inc., Naperville, Illinois
  - American Medical Research, Inc., Oak Brook, Illinois
  - Davis Clinic, Indianapolis, Indiana
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Pedia Research LLC, Owensboro, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Clinical Insights, Glen Burnie, Maryland
  - Neurocare, Inc., Newton, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Mid-Michigan Sleep Center, Grand Blanc, Michigan
  - Clinical Neurophysiology Services, P.C., Troy, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Synergy Clinical Research Center, Farmingdale, New York
  - Tristate Sleep Disorders Center, Cincinnati, Ohio
  - MD & Associates, Inc., Garfield Heights, Ohio
  - IPS Reserach Company, Oklahoma City, Oklahoma
  - Pahl Pharmaceutical Professionals, LLC, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Eminence Research, LLC, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Tulsa, Oklahoma
  - Paradigm Research Professional, LLP, Tulsa, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Carolina Clinical Trials Inc., Charleston, South Carolina
  - InSite Clinical Research LLC, DeSoto, Texas
  - Claghorn-Lesem Research Clinic, Houston, Texas
  - Allegiant Clinical Research, LLC, Houston, Texas
  - MD, Houston, Texas
  - Todd J. Swick, MD, PA, Houston, Texas
  - MD, Lubbock, Texas
  - The Mech Center, Plano, Texas
  - Aspen Clinical Research, LLC, Orem, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington

REFERENCES:
- [Derived] Sangal RB, Blumer JL, Lankford DA, Grinnell TA, Huang H. Eszopiclone for insomnia associated with attention-deficit/hyperactivity disorder. Pediatrics. 2014 Oct;134(4):e1095-103. doi: 10.1542/peds.2013-4221. PMID 25266438

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Numbers provided in any of the rows in the participant flow section are for subjects who were randomized. Number of participants in the Baseline Characteristics refers to only the subjects who were randomized AND had taken at least one dose of study drug during the doubleblind treatment period. Three subjects did not receive study medication.
Groups:
- Pooled High Dose Eszopiclone: 2 mg eszopiclone for 6-11 years, 3 mg eszopiclone for 12-17 years
- Pooled Low Dose Eszopiclone: 1 mg eszopiclone for 6-11 years, 2 mg for 12-17 years
Period: Overall Study
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Started | 162 | 163 | 161
Completed | 126 | 122 | 123
Not Completed | 36 | 41 | 38
Not completed — Adverse Event | 5 | 5 | 3
Not completed — Lost to Follow-up | 6 | 3 | 5
Not completed — Physician Decision | 0 | 3 | 1
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 13 | 16 | 15
Not completed — Other | 11 | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Pooled High Dose Eszopiclone: 2 mg eszopiclone for 6-11 years, 3 mg eszopiclone for 12-17 years once daily. This included only patients that were randomized (ITT population).
- Pooled Low Dose Eszopiclone: 1 mg eszopiclone for 6-11 years, 2 mg eszopiclone for 12-17 years once daily. This includes only patients that were randomized (ITT population).
- Placebo: Placebo Once Daily. This included only patients that were randomized (ITT population).
- Total: Total of all reporting groups
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo | Total
Number analyzed (Participants) | 160 | 163 | 160 | 483
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 160 | 163 | 160 | 483
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 00 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 11.3 (3.0) | 11.4 (3.0) | 11.6 (3.0) | 11.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 60 | 59 | 175
  Male | 104 | 103 | 101 | 308
Region of Enrollment [Number; unit: participants]
  United States | 160 | 163 | 160 | 483

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of the Double- Blind Treatment Period (Week 12) in Polysomnography (PSG) Defined Latency to Persistent Sleep (LPS).
Description: A central scoring facility was used to derive the PSG sleep parameters Latency to Persistent Sleep (LPS) from the epochs and stages collected via the PSG recordings. Each epoch is 30 seconds. The PSG parameters provided an objective assessment of the subject's sleep on a given night. Change from BL at Week 12 in LPS was derived from Week 12 LPS subtracted by BL LPS. Latency to persistent sleep (LPS; minutes): time from lights out to the first of 20 consecutive epochs (10 minutes) of non-wake, as determined by PSG recordings.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat (ITT) population with both baseline and week 12 LPS. ITT refers to only the subjects who were randomized AND had taken at least one dose of study drug during the doubleblind treatment period.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 123 | 122 | 121
minutes | -18.33 (3.91) | -23.45 (3.91) | -25.66 (3.92)
Statistical Analysis 1: Comparison: Pooled High Dose Eszopiclone vs Placebo; This endpoint was analyzed using ANCOVA with treatment group (pooled low dose eszopiclone, pooled high dose eszopiclone, and placebo) as a fixed effect and the baseline value as a covariate. Contrast statements were used to perform pairwise comparisons of the eszopiclone treatment groups to placebo. A Bonferroni adjustment was used for the 2 pairwise comparisons. Least squares means and the standard errors were presented for each treatment grou; Test type: Superiority or Other; p > 0.05, ANCOVA; Bonferroni adjustment was use for multiple comparisons; LS Mean Treatment Difference = 7.33, 97.5% CI 2-sided [-5.17 to 19.83], Standard Error of Mean 3.91 — Difference calculated as Eszopiclone minus placebo
Statistical Analysis 2: Comparison: Pooled Low Dose Eszopiclone vs Placebo; This endpoint was analyzed using ANCOVA with treatment group (pooled low dose eszopiclone, pooled high dose eszopiclone, and placebo) as a fixed effect and the baseline value as a covariate. Contrast statements were used to perform pairwise comparisons of the eszopiclone treatment groups to placebo. A Bonferroni adjustment was used for the 2 pairwise comparisons. Least squares means and the standard errors were presented for each treatment group; Test type: Superiority or Other; p > 0.05, ANCOVA; LS Mean Treatment Difference = 2.21, 97.5% CI 2-sided [-10.23 to 14.65], Standard Error of Mean 3.91

2. Secondary Outcome: Change From Baseline (Day 0) to Week 12 in PSG Defined Wake Time After Sleep Onset (WASO)
Description: A central scoring facility was used to derive the PSG sleep parameters Wake Time After Sleep Onset (WASO) from the epochs and stages collected via the PSG recordings. Each epoch is 30 seconds. The PSG parameters provided an objective assessment of the subject's sleep on a given night. Change from BL at Week 12 in WASO was derived from Week 12 WASO subtracted by BL WASO. Wake time after sleep onset (WASO; minutes): The number of wake epochs after the onset of persistent sleep to the end of the recording, divided by 2.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 WASO
Measure: Least Squares Mean (Standard Error); unit: Minutes
Groups:
- Placebo: Placebo 6-17 years once daily
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 123 | 122 | 121
Minutes | -23.35 (3.40) | -16.75 (3.41) | -17.30 (3.43)

3. Secondary Outcome: Change From Baseline in Clinical Global Improvement (CGI)-Parent/Caregiver at Week 12
Description: The CGI-I Parent/Caregiver was completed by the investigator based on interviews and interactions with the subject's parent or caregiver and represented their assessment of severity and improvement in the subject's symptoms since the start of the study. A 7 point scale was used for improvement with numeric values assigned to each of the responses: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), and very much worse (7).
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with Week 12 CGI Improvement from Parent/Caregiver
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 126 | 123 | 121
Units on a scale | 2.3 (0.1) | 2.6 (0.1) | 2.7 (0.1)

4. Secondary Outcome: Change From Baseline in CGI-Child at Week 12
Description: The CGI - I Child was completed by the investigator based on interviews and interactions with the subject and represented the subject's assessment of improvement in his/her symptoms since the start of the study. A 7 point scale was used for improvement with numeric values assigned to each of the responses: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), and very much worse (7).
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with Week 12 CGI Improvement from Child
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 126 | 123 | 121
Units on a scale | 2.3 (0.1) | 2.5 (0.1) | 2.7 (0.1)

5. Secondary Outcome: Change From Baseline (Day 0) to Week 12 in Conners' ADHD Inattention Rating Scale.
Description: The Conners' 3 -Parent Short Form was completed by the parent and provided an assessment of Attention-Deficit/ Hyperactivity Disorder (ADHD) and the most common comorbid problems and disorders in children and adolescents. It is a multi-informant assessment of children and adolescents between 6 and 18 years of age that took into account home, social and school settings. The short version of the Conners' 3 -Parent Short Form was a subset of items from the full-length form, and included the Conners' 3 Content Scales of Inattention, Hyperactivity/Impulsivity, Learning Problems, Executive Functioning, Aggression, and Peer/Family Relations. The scale scores were presented as standardized age and gender based t scores. Inattention score was used for this endpoint. The lowest scale score is 40 (best) and the highest is 90 (worse)].
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 Conners' ADHD Inattention rating scale
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 126 | 122 | 120
units on a scale | -8.8 (1.0) | -5.8 (1.0) | -7.1 (1.0)

6. Secondary Outcome: Change From Baseline to Week 12 in Subjective SL (Sleep Latency)
Description: A Sponsor produced sleep questionnaire asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of SL over a pre-defined time period. SL is subjective time to fall asleep.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 Subjective sleep latency
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 122 | 121 | 121
Minutes | 0.5 (1.1) | 0.6 (1.1) | 0.6 (1.1)

7. Secondary Outcome: Change From Baseline to Week 12 in Subjective Wake Time After Sleep Onset (WASO).
Description: A Sponsor produced sleep questionnaire asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of WASO over a pre-defined time period. WASO is the aggregate duration of awakenings from the time subjects fall asleep until last awakening. Wake time after sleep onset (WASO; minutes): The number of wake epochs after the onset of persistent sleep to the end of the recording, divided by 2.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 subjective WASO
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 122 | 122 | 120
Minutes | 0.2 (1.2) | 0.3 (1.2) | 0.3 (1.2)

8. Secondary Outcome: Change From Baseline to Week 12 in PSG Defined Sleep Efficiency (SE)
Description: A central scoring facility was used to derive the PSG sleep parameter of Sleep Efficiency (SE) from the epochs and stages collected via the PSG recordings. The PSG parameters provided an objective assessment of the subject's sleep on a given night. Sleep efficiency: (total sleep time)/(total recording time) x 100. For this endpoint, total sleep time was defined as the number of non-wake epochs from the beginning of recording to the end of recording divided by 2. If total recording time was greater than 960 epochs (480 minutes), total sleep time was calculated from the PSG truncated at 480 minutes.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 PSG defined sleep efficiency
Measure: Least Squares Mean (Standard Error); unit: percentage of SE
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 124 | 122 | 121
percentage of SE | 7.31 (1.07) | 7.40 (1.08) | 7.94 (1.08)

9. Secondary Outcome: Change From Baseline to Week 12 in PSG Defined Number of Awakenings After Sleep Onset (NAASO).
Description: A central scoring facility was used to derive the PSG sleep parameter of Number of Awakenings after Sleep Onset (NAASO). The PSG parameters provided an objective assessment of the subject's sleep on a given night. Number of awakenings: The number of times, after onset of persistent sleep, that there was a wake entry of at least one-minute duration. Each awakening must have been separated by an epoch of non rapid eye movement (NREM) sleep stage 2, 3/4, or rapid eye movement (REM) sleep.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 PSG defined of Awakenings After Sleep Onset
Measure: Least Squares Mean (Standard Error); unit: Number of Awakenings after sleep onse
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 123 | 122 | 121
Number of Awakenings after sleep onse | -2.0 (0.4) | -1.5 (0.4) | -0.7 (0.4)

10. Secondary Outcome: Change From Baseline to Week 12 in PSG Defined Total Sleep Time (TST)
Description: A central scoring facility was used to derive the PSG sleep parameter of Total Sleep Time (TST) from the epochs and stages collected via the PSG recordings. The PSG parameters provided an objective assessment of the subject's sleep on a given night. Total sleep time was defined as the number of non-wake epochs from the beginning of recording to the end of recording divided by 2. If total recording time was greater than 960 epochs (480 minutes), total sleep time was calculated from the PSG truncated at 480 minutes.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 PSG defined Total Sleep Time
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 124 | 122 | 121
Minutes | 36.90 (6.01) | 37.78 (6.05) | 35.38 (6.07)

11. Secondary Outcome: Change From Baseline to Week 12 in Subjective Total Sleep Time (TST).
Description: A Sponsor produced sleep questionnaire asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of TST over a pre-defined time period. TST is subjective total sleep time.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 subjective Total Sleep Time
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 121 | 123 | 122
Minutes | 77.2 (8.0) | 66.4 (8.0) | 49.2 (8.0)

12. Secondary Outcome: Change From Baseline to Week 11 in Subjective Sleep Latency (SL) Measured by Actigraphy Monitoring in the Actigraphy Population.
Description: A central scoring facility was used to derive the actigraphy sleep parameter of Sleep Latency (SL). Actigraphy data were used for additional efficacy evaluation as well as for the evaluation of rebound and withdrawal effects.
Time Frame: Baseline (Day 0) to Week 11
Population: The Actigraphy population included subjects in the ITT population for whom actigraphy data had been collected. All efficacy analyses of actigraphy data were performed using this population
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 85 | 83 | 98
Minutes | 0.90 (1.12) | 0.81 (1.12) | 0.93 (1.13)

13. Secondary Outcome: Change From Baseline to Week 11 in Subjective WASO From Actigraphy Population.
Description: A central scoring facility was used to derive the actigraphy sleep parameters Wake Time After Sleep Onset (WASO). Actigraphy data were used for additional efficacy evaluation as well as for the evaluation of rebound and withdrawal effects.
Time Frame: Baseline (Day 0) to Week 11
Population: Actigraphy population which included subjects in the ITT population for whom actigraphy data had been collected. All efficacy analyses of actigraphy data were performed using this population
Measure: Least Squares Mean (Standard Error); unit: Minutes
Groups:
- Pooled High Dose Eszopiclone: 2 mg eszopiclone for 6-11 years, 3 mg eszopiclone for 12-17 years once daily
- Pooled Low Dose Eszopiclone: 1 mg eszopiclone for 6-11 years, 2 mg eszopiclone for 12-17 years once daily
- Placebo: Placebo once daily
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 85 | 83 | 98
Minutes | 0.94 (1.06) | 1.02 (1.06) | 0.99 (1.07)

14. Secondary Outcome: Change From Baseline to Week 11 in Total Sleep Time (TST) Measured by Actigraphy Monitoring in the Actigraphy Population.
Description: A central scoring facility was used to derive the actigraphy sleep parameter of Total Sleep Time (TST). Actigraphy data were used for additional efficacy evaluation as well as for the evaluation of rebound and withdrawal effects.
Time Frame: Baseline (Day 0) to Week 11
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 85 | 83 | 98
Minutes | -4.72 (8.38) | 1.63 (8.28) | -6.02 (8.74)

15. Secondary Outcome: Change From Baseline to Week 12 in Pediatric Daytime Sleepiness Scale (PDSS) Total Score.
Description: The PDSS is a validated measure of excessive sleepiness specifically designed for use in school aged children. The scale allowed for measurement of sleepiness across several relatively sedentary activities and provided a means to unmask sleepiness that may not be recognized during more active situations. It consisted of 8 items that assessed the frequency of a sleep related behavior (eg, how often do you fall asleep or get drowsy during class periods; are you usually alert most of the day; how often do you think you need more sleep) using a 5-point Likert type scale (0 = never, 4 = always). All items were summed to obtain the PDSS total score. PDSS data were used for efficacy evaluation as well as for the evaluation of residual effects.The overall PDSS scores range from a low of 0 where the individual is endorsing each item at the lowest level of sleepiness to a high of 32 where the individual is endorsing each item at the highest level of sleepiness.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 in Pediatric Daytime Sleepiness Scale (PDSS) Total Score
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 126 | 120 | 121
units on a scale | -4.5 (0.5) | -4.0 (0.5) | -3.5 (0.5)

16. Secondary Outcome: Change From Baseline to Week 12 in Coding Copy Subtest / Digit Symbol Substitution Test (DSST) Scaled Score.
Description: These tests are standardized information processing tasks to assess recognition and recoding of sensory information. The subject was given 90 seconds to complete as many substitutions of symbols as possible according to a code provided on top of the sheet. The Coding Copy Subtest A was used for subjects 6-7 years of age and the Coding Copy Subtest B was used for subjects 8-16 years of age, and the DSST was used for subjects 17 years of age. The score is the number of squares filled in correctly. Individuals are measured against their own pre-treatment baseline to determine levels of impairment using the scaled score. Higher scores mean less impairment (or potentially improvement) as the number of correct substitutions generally improves as cognition improves. Scaled scores are used to account for age differences among test takers. Scaled scores range from 1 to 19, and higher scores indicate higher cognitive function.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 Coding Copy Subtest / Digit Symbol Substitution Test (DSST) Scaled Score
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 126 | 122 | 122
Score | 2.2 (3.3) | 2.1 (3.9) | 2.6 (5.3)

17. Secondary Outcome: Change From Baseline to Week 12 in Pediatric Quality-of-Life Scale (Short Form-10).
Description: The SF 10 Health Survey for Children is a 10 item care-giver completed assessment designed to measure children's health-related quality of life. The scale asked questions about the child's physical wellness, feelings, behavior, and activities at school and with family and friends. The SF 10 Physical and Psychosocial summary measures were scored such that higher scores indicated more favorable functioning.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 Pediatric Quality-of-Life Scale (Short Form-10)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 123 | 122 | 121
units on a scale
  Physical | 4.40 (0.64) | 3.07 (0.64) | 4.07 (0.65)
  Psychosocial | 2.234 (0.562) | 1.347 (0.566) | -0.121 (0.569)

18. Secondary Outcome: Change From Baseline to Week 12 in Subjective Number of Awakenings After Sleep Onset (NAASO).
Description: A Sponsor produced sleep questionnaire asked the subject or parent/guardian to report information about the subject's sleep and daytime functioning since the last visit. This questionnaire provided a subjective assessment of NAASO over a pre-defined time period.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population with both baseline and Week 12 Subjective Number of Awakenings After Sleep Onset (NAASO)
Measure: Least Squares Mean (Standard Error); unit: Number of Awakenings
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 123 | 122 | 122
Number of Awakenings | -1.1 (0.1) | -0.8 (0.1) | -1.0 (0.1)

19. Secondary Outcome: Change in School Tardiness/Attendance Reports at Week 12 (Days)
Description: School tardiness/attendance reports were to be collected when subject was actively enrolled in school (fall and spring semesters only; summer school, camps or other school attendance was not recorded.) The School Tardiness Report captured the number of days that the subject was tardy to school, had partial attendance at school or was completely absent from school. Data were collected for the 30-day period prior to Baseline, 6-week period prior to Week 6, 6-week period prior to Week 12.
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 160 | 163 | 160
Days
  Number of Days Tardy | -0.4 (0.1) | -0.2 (0.1) | -0.3 (0.1)
  Number of Days of Partial Attendance | 0.1 (0.1) | -0.2 (0.1) | -0.1 (0.1)
  Number of Days Absent | 0.0 (0.08) | -0.2 (1.2) | 0.3 (2.0)

20. Secondary Outcome: Change in School Tardiness/Attendance Reports at Week 12 (Hours)
Description: as for outcome 19
Time Frame: Baseline (Day 0) to Week 12
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Number analyzed (Participants) | 160 | 163 | 160
Hours | -0.10 (0.05) | -0.12 (0.05) | -0.12 (0.05)

ADVERSE EVENTS:
Description: Numbers provided in any of the rows in the participant flow section are for subjects who were randomized. Number of Participants at Risk in this adverse event section refers to the subjects who were randomized AND had taken at least one dose of study drug during the doubleblind treatment period.
Arm/Group | Pooled High Dose Eszopiclone | Pooled Low Dose Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 2/159 | 0/163 | 0/161
Other Adverse Events (participants affected / at risk) | 72/159 | 68/163 | 55/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled High Dose Eszopiclone (N=159) | Pooled Low Dose Eszopiclone (N=163) | Placebo (N=161)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled High Dose Eszopiclone (N=159) | Pooled Low Dose Eszopiclone (N=163) | Placebo (N=161)
Headache (Nervous system disorders) | 22 (34) | 19 (27) | 19 (33)
Dysgeusia (Nervous system disorders) | 22 (22) | 8 (8) | 2 (2)
Dizziness (Nervous system disorders) | 13 (20) | 6 (6) | 3 (3)
Somnolence (Nervous system disorders) | 6 (7) | 4 (4) | 3 (7)
Abdominal pain upper (Gastrointestinal disorders) | 8 (14) | 6 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5) | 10 (10) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (6) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (6)
Abdominal Discomfort (Gastrointestinal disorders) | 8 (8) | 4 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 4 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 13 (15) | 7 (7)
Nasopharyngitis (Infections and infestations) | 6 (6) | 9 (9) | 7 (9)
Paryngitis (Infections and infestations) | 0 (0) | 2 (2) | 4 (5)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (9) | 4 (4)
Pyrexia (General disorders) | 8 (9) | 4 (5) | 5 (6)
Irritability (General disorders) | 0 (0) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 4 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
Per protocol, study did not have PSG adaptation nights at baseline and contained one PSG assessment post randomization visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other